CLINICAL TRIAL: NCT03384485
Title: Prevalence of Lysosomal Hydrolase Alpha-glagtosidase Deficiency in Patients
Brief Title: Prevalence of Lysosomal Hydrolase Alpha-glagtosidase Deficiency in Patients With Antiphospholipid Syndrome.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, yair levy, head of department internal medicine E, Meir Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0255-17MMC
Record Dates: First submitted 2017-11-28; First posted 2017-12-27 (Actual); Last update posted 2017-12-27 (Actual); Status verified 2017-11

CONDITIONS: Antiphospholipid Syndrome
MeSH Terms: conditions — Antiphospholipid Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- antiphospholipid syndrome (Other): blood test in patients that diagnosed with antiphospholipid syndrome to diagnose Fabry's disease
  Interventions: Diagnostic Test: antiphospholipid syndrome

INTERVENTIONS:
Diagnostic Test: antiphospholipid syndrome — blood test for enzyme test,plasma and Lys-3-3 plasma

SUMMARY:
Fabry disease, an X-linked disorder of glycosphingolipids that is caused by mutations of the GLA gene that codes for α-galactosidase A, leads to dysfunction of many cell types and includes a systemic vasculopathy. As a result, patients have a markedly increased risk of developing ischemic stroke, small-fiber peripheral neuropathy, cardiac dysfunction and chronic kidney disease. Because this disease is a rare disease most of the time it is misdiagnosed, so in this study we will check out the Prevalence of lysosomal hydrolase alpha-glagtosidase deficiency ( Fabry disease) in patients with Antiphospholipid Syndrome.

DETAILED DESCRIPTION:
the investigators would like to assess the prevalence of Fabry in men and women aged 18-100 who were diagnosed with antiphospholipid syndrome in our departmental clinic in 2000-2017 It is very important to diagnose Fabri that then the treatment of patients can vary dramatically.

The study will include 100 adult patients (18-100) men and women. Testing for the Fabri test in men is an enzyme test and will be performed subject to their consent to sign informed consent. In the women, an enzyme test will be carried out, and the plasma Lys-3-3 plasma storage, as recommended in the recently published diagnostic algorithms, is examined. If diagnosed, a patient will be referred to a genetic institute for further genetic counseling

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Antiphospholipid syndrome.
* able to read and sign inform concent

Exclusion Criteria:

• Fabry disease.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2018-08-01 (Estimated); Study Completion 2018-10-01 (Estimated)

PRIMARY OUTCOMES:
Lys-3-3 plasma | an average of 1 year
  blood test to find the enzyme for Fabry's disease

CONTACTS AND LOCATIONS:
Overall Officials: Yair Levy, Principal Investigator — head of department internal medicin E
Locations (1):
- Meir Medical Center, Kfar Saba, Israel